CLINICAL TRIAL: NCT00875602
Title: Evaluation of EverOn™ - A Contact-Free System for Measuring Heart Rate, Respiratory Rate and Motion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: NO need
Sponsor: EarlySense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHW ES-MRK-PROT-6
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2012-10

CONDITIONS: Post Surgical Pat., Medical Pat., Resp. Failure, Car.Arrest, Death
Keywords: All hospitalized patients in a general Med/ Surg unit
MeSH Terms: conditions — Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): before-after (retrospective) and concurrent controls as comparators with a prospective intervention group
- Study unit (Active Comparator): Hospitalized patients in the study group will be continously monitored / supervised by the contact-free device
  Interventions: Device: EverOn (EarlySense) contactless monitoring device

INTERVENTIONS:
Device: EverOn (EarlySense) contactless monitoring device — Hospitalized patients on the study unit are monitored by a contactless device
  Arms: Study unit

SUMMARY:
Evaluation of continuous monitoring device on patients Risk during hospitalization and nurse satisfaction level.

DETAILED DESCRIPTION:
To assess the effects of continuous patient monitoring using a contactless monitor in a medical-surgical unit on transfers and length of stay at higher level of care units

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04

PRIMARY OUTCOMES:
Evidence of benefit to caregivers and patients | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Harvey V Brown, MD, Principal Investigator — CHW
Locations (1):
- CHMC, Los Angeles, California, United States